CLINICAL TRIAL: NCT06568055
Title: Investigation of Refractory CMV (Cytomegalovirus) Infection or Disease, After Kidney Transplantation, Using UK (United Kingdom) National Registry of Rare Kidney Diseases (RaDaR)
Brief Title: A Study of Cytomegalovirus (CMV) Infection After Kidney Transplant in Adults in the United Kingdom
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4012
Record Dates: First submitted 2024-08-09; First posted 2024-08-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cytomegalovirus (CMV)
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Refractory CMV group: Participants who had a kidney transplantation (including re-transplantation) with refractory CMV infection will be identified from five solid organ transplantation centres in England and followed retrospectively for at least 6 months and up to 7 years until the end of 2024 or exit date from the cohort for any reasons, including death or end of participation in the registry (follow up period).
  Interventions: Other: No Intervention
- Reference cohort of non-refractory CMV group: Participants with non-refractory CMV infection who have responded to initial anti-CMV therapy post-transplant with no CMV refractory to treatment will be followed retrospectively for at least 6 months and up to 7 years until the end of 2024 or exit date from the cohort for any reasons, including death or end of participation in the registry (follow up period).
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
This observational study intends to retrospectively gather information on cytomegalovirus (CMV) infection management in the United Kingdom (UK) over a period of 7 years (2017-2024). The main aims of this study are the following:

* To estimate the overall prevalence and annual rate of adults with refractory CMV infection after a kidney transplant and describe how such CMV infections are treated
* To describe how effective and well-tolerated the treatment was.
* To describe the demographic and clinical characteristics of adult participants with CMV infection (refractory and non-refractory).

In this study, already existing data will be reviewed and analysed from a UK database called the Registry of Rare Kidney Diseases (RaDaR) (NCT06065852). The study will only review data collected as part of routine clinical practice. The study will not impact the standard medical care and treatment of participants.

ELIGIBILITY:
Inclusion Criteria:

Refractory CMV group:

1. Participants aged greater than or equal to (>=) 18 years at index date
2. Kidney transplant recipients on or subsequent to June 2016.
3. CMV viraemia or disease identified as requiring treatment and which was refractory to previous CMV management (at least one course of therapy), with or without confirmed resistance.
4. At least six months follow up time (except for participants who have died earlier).

Reference cohort of non-refractory CMV group:

1. Participants aged >=18 years.
2. Kidney transplant recipients.
3. Received initial CMV management (at least one course of therapy).
4. At least six months follow up time (except for participants who have died earlier).

Exclusion Criteria:

Refractory CMV group:

1. Multi-organ transplant recipients.
2. Participation recorded in an anti-CMV prophylaxis or treatment clinical trial from 2010 onward.

Participants with non-refractory CMV are to be included as a reference to indicate impact of refractory CMV not responding to initial therapy on resource use and other outcomes.

Reference cohort of non-refractory CMV group:

1. Multi-organ transplant recipients.
2. Participation recorded in an anti-CMV prophylaxis or treatment clinical trial from 2010.
3. CMV viremia or disease refractory to any previous anti-CMV therapy.
4. Treatment for CMV viremia or disease refractory to initial therapy during the follow up period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with refractory CMV infection post-kidney transplant will be included. The reference cohort will include all participants identified to have responded to initial anti-CMV therapy post-transplant with no CMV which required the treatment of a 2nd anti-CMV agent during this episode of infection.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Non-Refractory and Refractory CMV Post-Kidney Transplant in 2024 | 1 year
Number of New Non-Refractory and Refractory CMV Cases per Year | 7 years
Percentage of Participants Given Prophylaxis at the Time of Kidney Transplant | At the time of kidney transplant (up to 7 years)
Distribution of Drugs Prescribed for Prophylaxis | Up to 7 years
Duration of Prophylactic Treatment | Up to 7 years
Dose of Prophylactic Treatment | Up to 7 years
Distribution of Drugs Prescribed for Initial Anti-CMV Treatment | Up to 7 years
Duration of Initial Anti-CMV Treatment | Up to 7 years
Dose of Initial Anti-CMV Treatment | Up to 7 years
Distribution of Drugs Prescribed as Anti-CMV Treatment Subsequent to Initial Therapy in Participants With Refractory CMV | Up to 7 years
  Distribution of drugs prescribed as anti-CMV treatment subsequent to initial therapy (that is, valganciclovir, ganciclovir, foscarnet, cidofovir, cytotect, maribavir) in participants with refractory CMV will be reported.
Duration of Time on Anti-CMV Treatment Subsequent to Initial Anti-CMV Therapy | Up to 7 years
Dose of Anti-CMV Treatment Subsequent to Initial Anti-CMV Therapy | Up to 7 years
Percentage of Participants With Refractory CMV Who Switched Type of Anti-CMV Treatment Subsequent to Initial Therapy in Six-Month Follow up Period | 6 months follow up period from index date
Time to Switch of Drug for Anti-CMV Treatment Subsequent to Initial Therapy | Up to 7 years
Number of Switches per Participants in Six-Month Follow up Period | 6 months follow up period
  The index date for all participants will be the earliest date between 1st January 2017 and 30th June 2024 when initial treatment for CMV was initiated.
Number of Participants as per Positioning of Marabivir in the Treatment Pathway | Up to 7 years
  Number of participants as per positioning of marabivir in the treatment pathway with first, second or third line of anti-CMV treatment subsequent to initial therapy will be reported.
Percentage of Participants With Viral Clearance During the Follow up Period | 6 months follow up period
  Viral clearance is defined as CMV concentration below detectable level.
Time to Viremia Recurrence From Documented Clearance or Cessation of Anti-CMV Treatment | Up to 7 years
Percentage of Participants With Recurrence of CMV Infection | Up to 7 years
Number of Hospital Admissions (per Year and Overall) | Up to 7 years
Reasons for Hospital Admission | Up to 7 years
Number of Hospitalisations (Including Intensive Care) per Participant in Six-Month Follow up Period | 6 months of follow up period
Duration of Hospitalisation | Up to 7 years
Number of Outpatient Visits in Six-month Follow up Period | 6 months of follow up period
Percentage of Participants With Graft Loss in Six-month Follow up Period | 6 months of follow up period from index date
Number of Occurrences of Each Reason for Graft Loss Listed in the Registry | Up to 7 years
  Graft loss being defined as re-establishment of long-term dialysis or estimated glomerular filtration rate (eGFR) of less than (<) 15 milliliter per minute (mL/min).
Percentage of Participants With Graft Loss Over Time for Refractory Versus non-Refractory Group | Up to 7 years
Number of Participants Who Died | Up to 7 years
Time to Death From Index Date/Transplant Date | From Index date/transplant date up to 7 years
  The index date for all participants will be the earliest date between 1st January 2017 and 30th June 2024 when initial treatment for CMV was initiated.
Number of Mortality (All-cause Death) | Up to 7 years
Number of Participants With Reasons for Mortality | Up to 7 years
Change in Renal Function (Estimated Glomerular Filtration Rate [eGFR]) From Index Date to Six-month Follow up | From index date to 6 months of follow up period
  The index date for all participants will be the earliest date between 1st January 2017 and 30th June 2024 when initial treatment for CMV was initiated.
Change in White Cell Count (Neutrophils) From Index Date to Six-month Follow up | From index date to 6 months of follow up period
  The index date for all participants will be the earliest date between 1st January 2017 and 30th June 2024 when initial treatment for CMV was initiated.
Percentage of Participants with Diabetes, Hypertension, and Cardiovascular Disease at the Time of Transplant | At the time of transplant (up to 7 years)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- RaDaR (part of the UK Kidney Association), Bristol, Southwestern England, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/5220278534c14c90??page=1&idFilter=TAK-620-4012